CLINICAL TRIAL: NCT03604263
Title: ArcticLine Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: MDT16015
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Results first posted 2020-05-20 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation; Atrial Flutter
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment Arm (Experimental): Subjects enrolled and treated with ArcticLine Cardiac Cryoablation Catheter
  Interventions: Device: ArcticLine Cardiac Cryoablation Catheter

INTERVENTIONS:
Device: ArcticLine Cardiac Cryoablation Catheter — Cryoablation
  Other Names: Arctic Front Advance Cardiac Cryoablation Catheter; Freezor MAX Cardiac Cryoablation Catheter; FlexCath Advance Steerable Sheath

SUMMARY:
The purpose of the ArcticLine Feasibility Study is to collect preliminary safety and effectiveness data on the ArcticLine Catheter.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of symptomatic persistent AF:

  * Defined as having a continuous episode that is sustained beyond 7 days documented via consecutive ECG recordings, or
  * Defined as having a continuous episode that is sustained beyond 7 days documented by an ECG recording and one doctor note indicating the patient had symptoms consistent with AF
* Age 18 through 80 years old
* Failure or intolerance of at least one Class I or III antiarrhythmic drug
* Subject is able and willing to consent to participate in the study and will commit to completion of all follow-up requirements

Exclusion Criteria:

* Longstanding persistent AF, defined as continuous AF greater than 12 month duration
* Left atrial diameter greater than 5.0 cm
* Active systemic infection
* History of thromboembolic event within the past 6 months or evidence of intracardiac thrombus at the time of the procedure
* Prior left atrial ablation attempt, with exception of:

  * Any pulmonary vein isolation attempt to treat AF, or
  * Successful ablation to treat Wolff-Parkinson White syndrome
* History of left atrial tachycardia
* History of cardiac ablation within 90 days of planned clinical study procedure
* Planned concomitant ventricular ablation
* Cryoglobulinemia
* Structural heart disease of clinical significance including:

  * NYHA Class IV Heart Failure
  * Diagnosed with NYHA Class III Heart Failure for more than six months at time of the study ablation procedure
  * LVEF less than 35%
  * Any cardiac surgery (e.g. CABG) within 3 months of the ablation procedure
  * Any mechanical heart valve, prior aortic or tricuspid valve replacement (e.g. valvotomy, valve replacement), or tricuspid valve repair
  * Severe mitral valve regurgitation or stenosis
  * Significant congenital anomaly or anatomy unable to accommodate device
* Prior surgical maze procedure
* Unstable angina
* Myocardial infarction within 3 months of the ablation procedure
* Presence of primum or secundum atrial septal defect
* Anomalous pulmonary venous return
* Prior surgery for congenital heart disease, including atrial septal defect repair
* Hypertrophic cardiomyopathy with LV septal wall thickness >1.5 cm
* Uncontrolled hyperthyroidism
* Thrombocytosis, thrombocytopenia (including history of heparin-induced thrombocytopenia)
* Severe comorbidity or poor general physical/mental health that, in the opinion of the investigator, will not allow the subject to be a good study candidate
* History of blood clotting or bleeding abnormalities
* Contraindication to all anticoagulation (e.g. novel oral anticoagulants, heparin or warfarin)
* Pregnant, nursing or planning to become pregnant during study duration
* Enrollment in another clinical trial without prior approval from Medtronic
* Presence or use of left atrial appendage closure device
* Presence of or planned implantation of a pacemaker, implantable cardiac defibrillator, implantable loop recorder or cardiac resynchronization device with permanent lead placement
* Pre-existing hemidiaphragmatic paralysis
* Life expectancy less than one year
* Known drug or alcohol dependency
* Existing pulmonary vein stent(s)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Pelosi, M.D., Principal Investigator — University of Michigan
Locations (4):
- United States (3):
  - BayCare Medical Group Cardiology, Tampa, Florida
  - University of Michigan, Ann Arbor, Michigan
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Arm
Started | 17
Completed | 15
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Baseline BMI [Mean (Standard Deviation); unit: kg/meter-squared] | 31.6 (4.6)
Baseline Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 145.1 (12.4)
Baseline Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 81.8 (12.2)
Heart Rate [Mean (Standard Deviation); unit: beats/min] | 74.7 (19.2)
LVEF (%) [Mean (Standard Deviation); unit: percentage of ejected blood] | 56.3 (8.1)
Left Atrial Diameter (mm) [Mean (Standard Deviation); unit: mm] | 44.7 (4.1)
NYHA Class [Count of Participants; unit: Participants] — NYHA is a heart failure classification system ranging from I (No limitations) to IV (Severe limitations). Class II indicates Mild symptoms and Class III indicates Marked symptoms.
  Participants
    Class I | 4
    Class II | 2
    Subject Does Not Have Heart Failure | 9
Time from Initial AF Diagnosis (months) [Mean (Standard Deviation); unit: months] | 97.6 (68.6)
Months of Continuous AF [Mean (Standard Deviation); unit: months] | 1.8 (1.7)
Time from First Documented Persistent AF [Mean (Standard Deviation); unit: months] | 18.7 (20.2)
Number of Failed AADs [Mean (Standard Deviation); unit: drugs] | 1.9 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Primary Safety Events With an Onset Date Within 7 Days Post-procedure.
Description: A primary safety event is defined as:
  An ArcticLine Catheter-related or ArcticLine cryoablation procedure-related SAE with an onset date within 7 days post-procedure (except as noted below), as adjudicated by the Clinical Events Committee (CEC), described as follows:
  * Atrioesophageal fistula*
    * Includes atrioesophageal fistula with an onset date at any time after the study cryoablation procedure and is adjudicated by the CEC as either ArcticLine Catheter-related or ArcticLine cryoablation procedure-related.
  * Cardiac perforation/tamponade
  * Cerebrovascular accident
  * Death
  * Esophageal injury
  * Major bleeding
  * Myocardial infarction
  * Pericarditis
  * Phrenic nerve injury (ongoing at hospital discharge)
  * Transient ischemic attack
  * Vagal nerve injury resulting in esophageal dysmotility or gastroparesis
  * Vascular access complications
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 15
Participants | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 1/15
Serious Adverse Events (participants affected / at risk) | 6/15
Other Adverse Events (participants affected / at risk) | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=15)
Atrial Fibrillation (Cardiac disorders) | 3 (3)
Anal Fissure (Gastrointestinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=15)
Atrial Fibrillation (Cardiac disorders) | 4 (5)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Anxiety Disorder (Psychiatric disorders) | 1 (1)
Atrial Flutter (Cardiac disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Chest Discomfort (General disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Gastrointestinal Disorder (Gastrointestinal disorders) | 1 (1)
Heart Rate Irregular (Investigations) | 1 (1)
Oedema Peripheral (General disorders) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Peripheral Swelling (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Ventricular Extrasystoles (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (5):
  • Study Protocol: CIP version 1.0 (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/63/NCT03604263/Prot_001.pdf
  • Study Protocol: CIP version 3.0 (2018-03-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT03604263/Prot_002.pdf
  • Study Protocol: CIP version 4.0 (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/63/NCT03604263/Prot_003.pdf
  • Study Protocol: CIP version 5.0 (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/63/NCT03604263/Prot_004.pdf
  • Statistical Analysis Plan (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/63/NCT03604263/SAP_000.pdf